CLINICAL TRIAL: NCT07252921
Title: A Phase II, Multicenter, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Efficacy and Safety of HRS-9190 for Injection as a Neuromuscular Blocking Agent for Tracheal Intubation During General Anesthesia Induction in Adult Patients Undergoing Elective Surgery
Brief Title: Safety and Efficacy of HRS-9190 Compared to Rocuronium for Tracheal Intubation in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9190-201
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: HRS-9190 (Experimental)
  Interventions: Drug: HRS-9190
- Treatment group B: HRS-9190 (Experimental)
  Interventions: Drug: HRS-9190
- Treatment group C: Rocuronium Bromide Injection. (Active Comparator)
  Interventions: Drug: HRS-9190

INTERVENTIONS:
Drug: HRS-9190 — HRS-9190; low dose
  Arms: Treatment group A: HRS-9190
Drug: HRS-9190 — HRS-9190; high dose
  Arms: Treatment group B: HRS-9190
Drug: HRS-9190 — Rocuronium Bromide Injection
  Arms: Treatment group C: Rocuronium Bromide Injection.

SUMMARY:
The study will enroll adult patients scheduled for elective surgery requiring general anesthesia with tracheal intubation. Participants will be randomly assigned to receive either HRS-9190 for Injection or Rocuronium. The primary objective is to assess the efficacy of HRS-9190 in providing adequate neuromuscular blockade for successful tracheal intubation. Secondary objectives include evaluating the onset time, duration of action, and recovery profile of neuromuscular blockade. Safety assessments will include monitoring of adverse events, vital signs, laboratory parameters, and other safety indicators throughout the study period. The hypothesis of this study is that HRS-9190 for Injection could provide effective neuromuscular relaxation for tracheal intubation, with a satisfied safety profile in the target patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia surgery
3. Meet specified age and body mass index (BMI) criteria
4. Conform to the ASA Physical Status Classification
5. Use of highly effective contraception for a specified period if applicable

Exclusion Criteria:

1. Scheduled for specific high-risk surgical procedures
2. History of significant neuromuscular, cardiovascular, respiratory, or neurological disorders
3. History of conditions affecting drug metabolism or anesthesia risk
4. Abnormal laboratory values indicating significant clinical abnormalities
5. Positive serology for specified infectious diseases
6. Known hypersensitivity to related medications
7. Recent use of medications interfering with neuromuscular function
8. History of mental illness, cognitive impairment, or epilepsy
9. Participation in another clinical trial within a specified period
10. Any other condition deemed unsuitable by the investigator
11. Pregnant or nursing women
12. Unwilling to use birth control during the specified period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-10-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Intubation conditions | Within 5 minutes after administration of the study drug
  Proportion of subjects with excellent or good intubation conditions as assessed by the Cooper score

SECONDARY OUTCOMES:
Time to Maximum Inhibition (Onset Time) | From start of study drug administration until the time when T1 reaches 0% (maximum suppression), Estimated within 5 minutes
  The time from the start of injection of the study drug to the time when T1 reaches 0% of its baseline value, indicating complete neuromuscular blockade and maximum drug effect.
Time to Successful Tracheal Intubation | From start of study drug administration to the completion of tracheal intubation, Estimated within 5 minutes
  The time from the start of injection of the study drug to the time when the endotracheal tube is correctly placed and secured, as confirmed by the anesthesiologist.
Time to Recovery of T1 to 10%/25% of Baseline | From start of study drug administration until the time when T1 recovers to 10% /25% of its baseline value, Estimated within 30 minutes
  The duration of action measured as the time from injection to the time when the first twitch (T1) recovers to 10%/25% of its pre-drug baseline height.
Time to Recovery of Train-of-Four Ratio (TOFr) to 0.4/0.7/0.9 | From start of study drug administration until the time when the TOFr recovers to 0.4/0.7/0.9, Estimated from 15 to 90 minutes
  The time from injection to recovery of the ratio of the fourth twitch (T4) to the first twitch (T1) to 0.4, which is a marker of adequate recovery for spontaneous ventilation.
Recovery Index (T1 25% to 75% and T1 5% to 95%) | within 2 hours after administration of research drug

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided